CLINICAL TRIAL: NCT05714293
Title: CT-evaluation of Coronary Ostia Height After Surgical Aortic Valve Replacement.
Acronym: CORONATE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5316
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Regurgitation, Aortic; Stenoses, Aortic; Aortic Regurgitation; Aortic Stenosis, Severe; Coronary; Obstruction; Valve Disease, Aortic
Keywords: Aortic valve replacement; Aortic valve bioprosthesis; Coronary ostia obstruction; Valve-in-valve; Transcatheter aortic valve implantation; Aortic valve stenosis; Tricuspid aortic valve; Aortic valve regurgitation; CT coronary angiogram; Transcatheter aortic valve replacement
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Bites and Stings; Aortic Valve Disease | interventions — Contrast Media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical Aortic Valve Replacement (Experimental): Patients undergoing surgical aortic valve replacement with a bioprosthesis will be asked to perform a thorax CT scan before surgery and one more at least 90 days after surgery.
  Interventions: Radiation: CT scan with contrast medium

INTERVENTIONS:
Radiation: CT scan with contrast medium — Multi-detector CT scan (if possible with prospective-ECG gated sequential scan) with contrast medium injection of nonionic contrast agent. All CT datasets will be analysed for the qualitative and quantitative assessment of the aortic root. The coronary height will be assessed at baseline in relation to the aortic annulus and in relation to the stent of the bioprostheses after aortic valve replacement.
  Other Names: CT scan

SUMMARY:
The goal of this interventional, single-center study is to demonstrate if there is a change in the coronary ostia height after surgical aortic valve replacement and if it depends on the type of prosthesis or surgical technique used. The study involves patients undergoing elective surgical aortic valve replacement with a bioprosthesis. Participants enrolled will undergo a CT scan before and after surgery (at least 90 days after surgery) to analyze coronary ostia height.

DETAILED DESCRIPTION:
Aortic valve stenosis is the most frequent heart valve disease in the adult population. The development of biological prostheses with slower valve degeneration and easier antithrombotic management and changes in the indications for the treatment of this valve disease, have allowed a reduction in the age in which such prostheses are implanted thus leading to a greater use of biological prostheses rather than mechanical ones. In the next few years this will cause a higher rate of structural valve degeneration resulting in stenosis and/or insufficiency. In patients considered to be at high surgical risk, the transcatheter implantation of a valve-in-valve (VIV) represents a valid alternative to standard surgery, except for coronary obstruction which appears more frequent in VIV procedures, especially in patients receiving VIV after surgical aortic valve replacement. The risk factors mainly associated with this complication are represented by the type of implanted prostheses and the anatomical relationship between the coronary ostia and the expected final position of the cusps of the bioprostheses transcatheter-implanted.Recent studies have demonstrated how coronary height seems to be significantly reduced in case of surgical aortic valve replacement with a supra-annular technique, as occurs in our center.

Aim of this interventional, single-center study is to demonstrate whether there is a change in the coronary ostia height after surgical aortic valve replacement and whether it possibly depends on the type of prosthesis.

All patients undergoing elective aortic valve replacement surgery at our institution who meet the inclusion criteria for the study will be contacted to perform a postoperative CT scan at least 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Aortic valve stenosis or insufficiency with indication for elective aortic valve replacement with a bioprosthesis;
* Possible concomitant coronary artery disease with indication for surgical or percutaneous revascularization;
* CT imaging of the thorax with iodinated contrast agent carried out before surgery;
* Signed informed consent, inclusive of release of medical information.

Exclusion Criteria:

* Aortic valve replacement in bicuspid valve or endocarditis;
* Aortic valve replacement associated with surgery of ascending aorta/aortic root;
* Aortic valve replacement associated with other cardiac valve surgery;
* Previous cardiac surgery of any kind;
* Patient unable to give informed consent or potentially noncompliant with the study protocol, in the judgment of the investigator;
* Participation in another clinical trial that could interfere with the endpoints of this study;
* Pregnant at time of screening;
* Allergy or hypersensitivity to iodinated contrast agent;
* End-stage renal disease on dialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Coronary ostia height differences. | At least 90 days after surgery
  Differences in coronary ostia height before and after surgical aortic valve replacement.

SECONDARY OUTCOMES:
Coronary ostia height differences between different bioprostheses. | At least 90 days after surgery
  Differences in coronary ostia height before and after surgical aortic valve replacement according to different bioprostheses used.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Massetti, MD, Principal Investigator — Policlinico Agostino Gemelli
Locations (1):
- Policlinico Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart BF, Siscovick D, Lind BK, Gardin JM, Gottdiener JS, Smith VE, Kitzman DW, Otto CM. Clinical factors associated with calcific aortic valve disease. Cardiovascular Health Study. J Am Coll Cardiol. 1997 Mar 1;29(3):630-4. doi: 10.1016/s0735-1097(96)00563-3. PMID 9060903
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Dunning J, Gao H, Chambers J, Moat N, Murphy G, Pagano D, Ray S, Roxburgh J, Bridgewater B. Aortic valve surgery: marked increases in volume and significant decreases in mechanical valve use--an analysis of 41,227 patients over 5 years from the Society for Cardiothoracic Surgery in Great Britain and Ireland National database. J Thorac Cardiovasc Surg. 2011 Oct;142(4):776-782.e3. doi: 10.1016/j.jtcvs.2011.04.048. PMID 21924147
- [Background] Capodanno D, Petronio AS, Prendergast B, Eltchaninoff H, Vahanian A, Modine T, Lancellotti P, Sondergaard L, Ludman PF, Tamburino C, Piazza N, Hancock J, Mehilli J, Byrne RA, Baumbach A, Kappetein AP, Windecker S, Bax J, Haude M. Standardized definitions of structural deterioration and valve failure in assessing long-term durability of transcatheter and surgical aortic bioprosthetic valves: a consensus statement from the European Association of Percutaneous Cardiovascular Interventions (EAPCI) endorsed by the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2017 Sep 1;52(3):408-417. doi: 10.1093/ejcts/ezx244. No abstract available. PMID 28874031
- [Background] Giordana F, Bruno F, Conrotto F, Saglietto A, D'Ascenzo F, Grosso Marra W, Dvir D, Webb J, D'Onofrio A, Camboni D, Grubitzsch H, Duncan A, Kaneko T, Toggweiler S, Latib A, Nerla R, Salizzoni S, La Torre M, Trompeo A, D'Amico M, Rinaldi M, De Ferrari G. Incidence, predictors and outcomes of valve-in-valve TAVI: A systematic review and meta-analysis. Int J Cardiol. 2020 Oct 1;316:64-69. doi: 10.1016/j.ijcard.2020.05.058. Epub 2020 May 26. PMID 32470529
- [Background] Bernardi FLM, Dvir D, Rodes-Cabau J, Ribeiro HB. Valve-in-Valve Challenges: How to Avoid Coronary Obstruction. Front Cardiovasc Med. 2019 Aug 23;6:120. doi: 10.3389/fcvm.2019.00120. eCollection 2019. PMID 31508426
- [Background] Coti I, Maierhofer U, Rath C, Werner P, Loewe C, Kocher A, Laufer G, Andreas M. Effect of conventional and rapid-deployment aortic valve replacement on the distance from the aortic annulus to coronary arteries. Interact Cardiovasc Thorac Surg. 2021 Jan 22;32(2):196-203. doi: 10.1093/icvts/ivaa247. PMID 33236042
- [Background] Bruno P, Cammertoni F, Rosenhek R, Mazza A, Pavone N, Iafrancesco M, Nesta M, Chiariello GA, Spalletta C, Graziano G, Sanesi V, D'Errico D, Massetti M. Improved Patient Recovery With Minimally Invasive Aortic Valve Surgery: A Propensity-Matched Study. Innovations (Phila). 2019 Oct;14(5):419-427. doi: 10.1177/1556984519868715. Epub 2019 Aug 21. PMID 31431105
- [Background] Freeman LA, Young PM, Foley TA, Williamson EE, Bruce CJ, Greason KL. CT and MRI assessment of the aortic root and ascending aorta. AJR Am J Roentgenol. 2013 Jun;200(6):W581-92. doi: 10.2214/AJR.12.9531. PMID 23701088
- [Background] Salgado RA, Leipsic JA, Shivalkar B, Ardies L, Van Herck PL, Op de Beeck BJ, Vrints C, Rodrigus I, Parizel PM, Bosmans J. Preprocedural CT evaluation of transcatheter aortic valve replacement: what the radiologist needs to know. Radiographics. 2014 Oct;34(6):1491-514. doi: 10.1148/rg.346125076. PMID 25310413
- [Background] Salemi A, Worku BM. Standard imaging techniques in transcatheter aortic valve replacement. J Thorac Dis. 2017 Apr;9(Suppl 4):S289-S298. doi: 10.21037/jtd.2017.03.114. PMID 28540072